CLINICAL TRIAL: NCT00560742
Title: Efficacy of the Mode of Delivery of Autologous Bone Marrow Cells Into Heart Scar Muscle for the Recovery of Contractile Function
Brief Title: Efficacy Study of Intramuscular or Intracoronary Injection of Autologous Bone Marrow Cells to Treat Scarred Myocardium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospitals, Leicester (Other)
Collaborators: British Heart Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PG04050; UHL ref: 7638
Record Dates: First submitted 2007-11-16; First posted 2007-11-20 (Estimated); Last update posted 2007-11-20 (Estimated); Status verified 2007-11

CONDITIONS: Myocardial Infarct; Bone Marrow Cells
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Control (Active Comparator)
  Interventions: Procedure: Control
- Intramuscular (Experimental)
  Interventions: Procedure: Intramuscular administration of bone marrow cells
- Intracoronary (Experimental)
  Interventions: Procedure: Intracoronary administration of bone marrow cells

INTERVENTIONS:
Procedure: Control — Coronary artery bypass grafting without bone marrow cells injection
  Arms: Control
Procedure: Intramuscular administration of bone marrow cells — Coronary artery bypass grafting, and intramuscular administration of bone marrow cells into myocardial scar
  Arms: Intramuscular
Procedure: Intracoronary administration of bone marrow cells — Coronary artery bypass grafting, and intracoronary administration of bone marrow cells into myocardial scar
  Arms: Intracoronary

SUMMARY:
The purpose of this study is to determine whether the administration of patient's own bone marrow cells into scar areas of the heart, can improve the contractile function of these areas.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective CABG
* chronic irreversible myocardial scar
* coronary vessel supplying the scar must be amenable to bypass grafting

Exclusion Criteria:

* significant valvular heart diseases
* major organ failures, eg. heart, liver, renal etc
* pre-existing bone marrow conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2002-11; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Contractile function of treated scar areas | 6 months

SECONDARY OUTCOMES:
Global left ventricular functions | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Galiñanes, MD PhD FRCS, Principal Investigator — University Hospitals, Leicester
Locations (1):
- University Hospitals Leicester, Leicester, Leicestershire, United Kingdom